CLINICAL TRIAL: NCT01427569
Title: A Randomized, Placebo-controlled, Double-blind Phase II Study to Evaluate the Efficacy of IZN-6D4 Gel for the Treatment of Diabetic Foot Ulcers
Brief Title: Efficacy Study of IZN-6D4 Gel for the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Izun Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IWH-DFU-101-IL
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Chronic wound
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IZN-6D4 Gel (Experimental): patients in this arm will be treated by twice a week bandaging the wound with active IZN-6D4 Gel
  Interventions: Drug: IZN-6D4 Gel
- Placebo Hydrogel (Placebo Comparator): patients in this arm will be treated by twice a week bandaging the wound with a hydrogel used for wound care, but without the active IZN-6D4
  Interventions: Other: Placebo hydrogel

INTERVENTIONS:
Drug: IZN-6D4 Gel — Standard wound therapy plus twice weekly topical application of hydrogel containing botanical extracts.
  Other Names: Curasite
  Arms: IZN-6D4 Gel
Other: Placebo hydrogel — Standard wound therapy plus twice weekly topical application of color-matched placebo hydrogel
  Other Names: Teva Gel
  Arms: Placebo Hydrogel

SUMMARY:
The purpose of this study is to determine if topical application of a hydrogel that contains plant extracts will improve healing of diabetic foot ulcers when compared to treatment with a hydrogel alone.

DETAILED DESCRIPTION:
This is a multi center, double-blind, randomized, placebo-controlled trial. A total of 80 patients will be randomized according to a 1: 1 randomization schedule. To participate in the trial, patients must have a current Diabetic Foot Ulcer (DFU) for between 60 days to 2 years at the screening visit. In the 2-week period between screening and baseline visit, the patient's DFU must not have healed by 30% or more, in wound area, while being treated with SWT twice a week during this screening period.

During the treatment period of 4 weeks all patients will be examined on a weekly basis by the site staff. Treatment with SWT plus the study gel (IZN-6D4 Gel or placebo gel) (including any necessary debridement) will be administered at these weekly visits. In addition, the patient or caregiver will be trained to perform SWT plus the study treatment at home once midweek between visits.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of diabetes mellitus type 1 or 2
* Foot ulcer Wagner grade 1 or 2
* Ulcer between 1 square cm and 8 square cm present for at least 60 days and not more than two years
* HgbA1C less than 10%
* Able to comply with all procedures

Exclusion Criteria:

* Wound area decrease of greater than 30% between screening and baseline visits
* Gangrene on any part of the affected foot
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The percent reduction in wound area at week 4 compared to the baseline visit | Weekly measurements of wound area from study initiation and through week 4

SECONDARY OUTCOMES:
The percent conversion of the wound bed to granulation tissue by week 4 compared to baseline | Weekly assessments from baseline through week 4
The percentage of lesions that demonstrate at least 40% reduction in area by the end of week 4 compared to baseline visit | Weekly assessments of wound area through week 4
The percentage of lesions that demonstrate at least 50% reduction in area by the end of week 4 compared to baseline visit | Weekly assessments of wound area from baseline through week 4

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Nussbaum, PhD, MD,, Study Director — Izun Pharma Ltd
Locations (1):
- Wolfson Medical Center, Holon, Israel